CLINICAL TRIAL: NCT01180517
Title: The Paclitaxel-Eluting PTCA-Balloon Catheter for the Treatment of Coronary Bifurcations
Brief Title: The Paclitaxel-Eluting Percutaneous Coronary Angioplasty (PTCA)-Balloon Catheter for the Treatment of Coronary Bifurcations
Acronym: PEPCAD-BIF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ralf Degenhardt, PhD (Other)
Collaborators: B. Braun Melsungen AG (Industry)
Responsible Party: Sponsor-Investigator, Ralf Degenhardt, PhD, Data Manager, Heart Centre Rotenburg
Organization: Heart Centre Rotenburg (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAG-G-H-1003
Record Dates: First submitted 2010-08-09; First posted 2010-08-12 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Angioplasty
Keywords: Angioplasty Balloon
MeSH Terms: interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug Eluting Balloon (Active Comparator)
  Interventions: Procedure: Percutaneous coronary intervention (PCI)
- Plain Old Balloon Angioplasty (POBA) (Active Comparator)
  Interventions: Procedure: PCI

INTERVENTIONS:
Procedure: Percutaneous coronary intervention (PCI) — balloon angioplasty
  Arms: Drug Eluting Balloon
Procedure: PCI — balloon angioplasty
  Arms: Plain Old Balloon Angioplasty (POBA)

SUMMARY:
The intention of this trial is to assess the safety and efficacy of Drug Eluting Balloon (DEB) application (SeQuent Please) to the side branch in percutaneous coronary intervention (PCI) of Medina 0,0,1 coronary bifurcation lesions. Patients will be randomized to treatment with Plain Old Balloon Angioplasty (POBA)or treatment with DEB.

ELIGIBILITY:
Inclusion Criteria (main):

* De-novo Medina type 0,0,1 bifurcational native coronary artery lesion (reference diameter:>2.0 mm <3.5 mm, length of stenosis: ≤ 10 mm), the diameter of the side branch shall be smaller or equal to the diameter of the distal end vessel

Exclusion Criteria (main):

* Reference side branch diameter > 3.5 mm
* Evidence of extensive thrombosis within target vessel
* Patients with another coronary stent implanted previously into the target branch or bifurcation ≤ 15 mm distant to the current lesion, drug eluting stents less than 9 months and bare metal stents or stents with passive coatings less than 3 months before the PEPCAD- BIF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-11; Primary Completion 2014-11 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
In-segment late lumen loss in the side branch at 9 months | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: F. X. Kleber, MD, Principal Investigator — Klinikum Ernst von Bergmann Potsdam, Germany
Locations (2):
- Germany (2):
  - Herzzentrum Dresden, Dresden
  - Klinikum Ernst von Bergmann, Potsdam